CLINICAL TRIAL: NCT03367299
Title: National Treatment Program With Sequential Chemotherapy and Blinatumomab to Improve Minimal Residual Disease Response and Survival in Philadelphia Chromosome-Negative B-Cell Precursor Adult Acute Lymphoblastic Leukemia
Brief Title: Sequential Chemotherapy and Blinatumomab to Improve MRD Response and Survival in Acute Lymphoblastic Leukemia
Acronym: LAL2317
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL2317
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Acute Lymphoid Leukemia; Philadelphia Chromosome-Negative B-Cell Precursor
Keywords: Acute Lymphoid Leukemia; Philadelphia Chromosome-Negative B-Cell Precursor; Adults; Minimal residual disease; Blinatumomab
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — Drug Therapy; blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Chemotherapy + Blinatumomab (Experimental): Treatment sequence consists of eight chemotherapy courses and two blinatumomab courses. Patients not in CR after chemotherapy course 2 will go off-study.
  Interventions: Drug: Chemotherapy + Blinatumomab

INTERVENTIONS:
Drug: Chemotherapy + Blinatumomab — Chemotherapy cycles are administered at 21-28 days intervals and each blinatumomab course is 28-day long.

SUMMARY:
The present study aims at analyzing the response to treatment of adult patients homogeneously treated with supportive care, chemotherapy and blinatumomab.

DETAILED DESCRIPTION:
Eligible patients with CD19+ Ph- BCP ALL (Philadelphia-negative B-cell precursor acute lymphoblastic leukemia) will receive homogeneous supportive care, chemotherapy and blinatumomab immunotherapy, and will be homogeneously analyzed for response at prefixed time points from induction day 1. For risk-oriented therapy, patients in complete remission (CR) will be stratified by risk class according to the diagnostic characteristics and MRD (minimal residual disease) study results during early consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent according to ICH/EU/GCP and national local laws.
* Age 18-65 years.
* A diagnosis of untreated Ph- CD19+ BCP ALL is required, either de novo or secondary to chemo-radiotherapy for another cancer. Pre-treatment with low-dose corticosteroids in patients presenting with hyperleukocytosis is allowed. Before enrolment and pre-phase is allowed only in patients presenting with severe, potentially life-threatening disease-related clinical symptoms. All diagnostic procedures need to be performed on freshly obtained bone marrow (BM) and peripheral blood (PB) samples.
* Full cytological, cytochemical, immunophenotypic, cytogenetic and molecular disease characterization according to the EGIL and WHO classifications.
* BM and PB sampling for MRD evaluations study. Detailed indications on patient registration, storage of representative diagnostic material and diagnostic work-up, including the shipping of samples for the diagnostic work-up and MRD follow-up studies are given in Appendix A.
* An ECOG performance status 0-2, unless a performance of 3 is unequivocally caused by the disease itself, (and not by pre-existing comorbidities,) and is considered and/or documented to be reversible following the application of anti-leukemic therapy and appropriate supportive measures.

Exclusion Criteria:

* Diagnosis of Burkitt's leukemia/lymphoma, CD19- BCP ALL, Ph+ ALL, T-ALL, lymphoblastic lymphoma (BM involvement by blast cells <25%).
* Active CNS leukemia documented by diagnostic lumbar puncture on days -1 to -5 prior to the first blinatumomab administration, or any other clinical sign or symptom ascribable to symptomatic/documented CNS disease at time of each planned blinatumomab course.
* Down's syndrome.
* A pre-existing, uncontrolled pathology such as heart failure (congestive/ischemic, acute myocardial infarction within the past 3 months, untreatable arrhythmias, NYHA classes III and IV), severe liver disease with serum bilirubin >3 mg/dL and/or ALT >3 x upper normal limit (unless attributable to ALL), kidney function impairment with serum creatinine >2 mg/dL (unless attributable to ALL), and severe neuropsychiatric disorder that impairs the patient's ability to understand and sign the informed consent, or to cope with the intended treatment plan. N.B. For altered liver and kidney function tests, eligibility criteria can be reassessed at 24-96 hours, following the institution of adequate supportive measures.
* Presence of serious, active, uncontrolled infections.
* Pre-existing HIV positive serology (i.e. already known before enrolment). If HIV positivity is detected after enrolment, the patient is put off study.
* A history of cancer that is not in a remission phase following surgery and/or radiotherapy and/or chemotherapy, with a life expectancy <1 year.
* Pregnancy declared by the patient, unless a decision is taken with the patient to induce a therapeutic abortion in order to carry on with the ALL therapy. A pregnancy test is performed at diagnosis, but does not preclude the enrolment into study. Fertile patients will be advised to adopt contraceptive methods while on treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Number of patients that obtain a negative Minimal Residual Disease (MRD) | At week 14 from study entry

SECONDARY OUTCOMES:
Number of patients in complete remission (CR) | At 32 months from study entry
Number of patients that reach disease-free survial | At 32 months from study entry
Number of patients that relapse | At 32 months from study entry
Number of patients that dye due to treatment | At 32 months from study entry
  Treatment-related mortality
Number of serious adverse events | At 32 months from study entry
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Renato Bassan, Study Chair — Azienda ULSS 12 "Veneziana" U.O. Ematologia Direttore Renato Bassan; Roberto Foà, Study Director — Policlinico Umberto I, Hematology Department.; Alessandro Rambaldi, Study Director — Ospedale di Bergamo
Locations (62):
- Italy (62):
  - AOU Ospedali Riuniti Umberto I - G.M. LANCISI - G. SALESI, Ancona
  - U.O.C. Ematologia e Terapia Cellulare - Ospedale "C. e G. Mazzoni" di Ascoli Piceno, Ascoli Piceno
  - Az.Ospedaliera S.G.Moscati, Avellino
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - UOC di Ematologia - Istituto Tumori - Giovanni Paolo II, Bari
  - UOC Ematologia Ospedale " Monsignor Raffaele Dimiccoli", Barletta
  - Azienda Ospedaliera - Papa Giovanni XXIII, Bergamo
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Policlinico S. Orsola - Malpighi, Bologna
  - Comprensorio Sanitario di Bolzano - Azienda Sanitaria dell'Alto Adige - Ematologia e Centro TMO - Ospedale S.Maurizio, Bolzano
  - Spedali Civili - Brescia - Azienda Ospedaliera - U.O. Ematologia, Brescia
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - S.C. Ematologia ASO S. Croce e Carle, Cuneo
  - Unità di Ricerca e di Malattie del sangue - Ematologia San Luca Vecchio, Florence
  - IRCCS_AOU San Martino-IST-Ematologia 1-Monoblocco 11°piano- lato ponente, Genova
  - UOC di Ematologia con trapianto Ospedale S. Maria Goretti, Latina
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - A.O.U. - Policlinico G. Martino Messina Oncologia Medica - U.O.C. Ematologia, Messina
  - U.O. di Ematologia- Ospedale dell'Angelo - Mestre, Mestre
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia, Milan
  - Ospedale Niguarda " Ca Granda" - SC Ematologia, Milan
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - S.C.D.U. Ematologia - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - U.O. CTMO Ematologia - Osp. S.Francesco, Nuoro
  - S.C.D.U.Medicina Interna a indirizzo ematologico, Orbassano
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - Oncoematologia -plesso ospedaliero "A. Tortora" di Pagani, Pagani
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - U.O. di Ematologia con trapianto - Centro di Riferimento Regionale per le coagulopatie rare nel bambino e nell'adulto - A.U. Policlinico "Paolo Giaccone", Palermo
  - Day Hospital dell'U.O.C di Ematologia e CTMO Padiglione 1, Parma
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della Misericordia, Perugia
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - U.O. Ematologia - AUSL Ospedale G. da Saliceto, Piacenza
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Ospedale "Infermi", Rimini
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza II Facoltà di Medicina e Chirurgia, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Padiglione Cesalpino - I piano - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S. Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Sezione di Ematologia Cancer Center Humanitas, Rozzano
  - UOC di Ematologia - AOU San Giovanni di Dio e Ruggi D'Aragona, Salerno
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia - A.O. Senese - Policlinico " Le Scotte", Siena
  - U.O.C. di Ematologia - A.O. " SS Annunziata" - P.O. S.G. Moscati, Taranto
  - Divisione di Ematologia dell'Università di Torino - "Città della Salute e della Scienza", Torino
  - Ematologia e Terapie Cellulari- A.S.O. Ordine Mauriziano, P.O. Umberto I-Ospedale, Torino
  - S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Struttura Complessa Ematologia - Azienda Ospedaliera Universitaria Integrata-Ospedale Maggiore, Trieste
  - Clinica Ematologica-Centro Trapianti e Terapie cellulari AOU,, Udine
  - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona
  - ULSS N.6 Osp. S. Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bassan R, Chiaretti S, Della Starza I, Santoro A, Spinelli O, Tosi M, Elia L, Cardinali D, De Propris MS, Piccini M, Lussana F, Annunziata M, Chiusolo P, Zappasodi P, Borlenghi E, Leoncin M, Califano C, Bocchia M, Di Raimondo F, Grimaldi F, Tiribelli M, Candoni A, Lico A, Audisio E, Lunghi M, Mianulli AM, Di Trani M, Arena V, Messina M, Piciocchi A, Fazi P, Rambaldi A, Foa R. Up-front blinatumomab improves MRD clearance and outcome in adult Ph- B-lineage ALL: the GIMEMA LAL2317 phase 2 study. Blood. 2025 May 22;145(21):2447-2459. doi: 10.1182/blood.2024027500. PMID 40009490
- See also: GIMEMA Foundation website — http://www.gimema.it